CLINICAL TRIAL: NCT03725657
Title: Using a Wrist-worn Accelerometer to Find a Correlation Between Exercise, Glycaemia and Insulin Dose in Type 1 Pediatric Patients, During a Camp: inCamp Study
Brief Title: Correlation Between Exercise and Insulin Dose in a Camp for Pediatric Type 1 Patients
Acronym: inCamp
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Angela Zanfardino, Principal Investigator, University of Campania Luigi Vanvitelli
Other Study IDs: inCamp1
Record Dates: First submitted 2018-10-28; First posted 2018-10-31 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Type1 Diabetes Mellitus; Hypoglycemia; Exercise
MeSH Terms: conditions — Hypoglycemia; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric: Pediatric Type1 Diabetes Mellitus patients

SUMMARY:
Intense exercise is a major challenge to the management of type 1 diabetes. The management is even more difficult, during a camp, probably due to increased hypoglycemia maybe from increase of intensity of physical activity.

The investigators want to evaluate steps, energy expenditure, sleep time and glycemic control and insulin dosage, through use of a wrist accelerometer, in pediatric type 1 patients attending a camp. Finding a correlation between these parameters could be useful not only for educational purposes but also in the development of algorithms for artificial pancreas.

DETAILED DESCRIPTION:
Background and Aims Intense exercise is a major challenge to the management of type 1 diabetes. The management is even more difficult, during a camp, probably due to increased hypoglycemia maybe from increase of intensity of physical activity. Few studies confirm this hypothesis but none evaluated the correlation between steps, energy expenditure, sleep time and glycemic control and insulin dosage.

Methods and Materials 60 patients with type 1 diabetes, aged 10 to 12 years, in multiinjection insulin therapy observed for 21 days (one week of camp, one week before and one after it). Food program was the same both at home and during the camp. They checked glycemia almost 5 times a day. A wrist accelerometer was used to evaluate sleep, steps and energy expenditure.

All data were recorded in a daily diary.

ELIGIBILITY:
Inclusion Criteria:

* diabetes onset > 1 year, multiple injection insulin therapy

Exclusion Criteria:

* Physical impossibility to movement, food allergy

Ages: 10 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: Pediatric Type1Diabetes patients
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

PRIMARY OUTCOMES:
Measure of steps through wrist accelerometer | three weeks
  number of steps
Measure of energy expenditure through wrist accelerometer | three weeks
  kcal
Measure of sleep expenditure through wrist accelerometer | three weeks
  hours of sleep

SECONDARY OUTCOMES:
Measure of glycemic control through glucometer | three weeks
  mmol/L
Measure of insulin dosage | three weeks
  Units/kg

CONTACTS AND LOCATIONS:
Locations (1):
- Centro di Diabetologia Pediatrica "G.Stoppoloni", Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Miller AR, Nebesio TD, DiMeglio LA. Insulin dose changes in children attending a residential diabetes camp. Diabet Med. 2011 Apr;28(4):480-6. doi: 10.1111/j.1464-5491.2010.03220.x. PMID 21204959
- [Result] Kelly D, Hamilton JK, Riddell MC. Blood glucose levels and performance in a sports cAMP for adolescents with type 1 diabetes mellitus: a field study. Int J Pediatr. 2010;2010:216167. doi: 10.1155/2010/216167. Epub 2010 Aug 2. PMID 20811595
- [Result] Bunn JA, Navalta JW, Fountaine CJ, Reece JD. Current State of Commercial Wearable Technology in Physical Activity Monitoring 2015-2017. Int J Exerc Sci. 2018 Jan 2;11(7):503-515. doi: 10.70252/NJQX2719. eCollection 2018. PMID 29541338